CLINICAL TRIAL: NCT02135939
Title: Effects of a Whole-food Plant-based Vegan Diet on Markers of Inflammation and Glucometabolic Profile in Patients With Coronary Artery Disease
Brief Title: Vegan vs AHA Diet on Inflammation and Glucometabolic Profile in Patients With CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-00292
Record Dates: First submitted 2014-05-07; First posted 2014-05-12 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease; Inflammation
MeSH Terms: conditions — Coronary Artery Disease; Inflammation | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- American Heart Association diet (Active Comparator): Participants randomized into this arm will follow an American Heart Association diet plan for 8 weeks.
  Interventions: Behavioral: Diet
- Whole-food plant-based vegan diet (Experimental): Participants randomized into this arm will be asked to follow a whole-food plant-based vegan diet plan for 8 weeks.
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Diet — Whole foods plant based vegan diet vs the American Heart Association-recommended diet
  Other Names: Vegan vs AHA-recommended diet

SUMMARY:
In this randomized study the investigators aim to determine the effects of a whole-food plant-based vegan diet on markers of inflammation and glucometabolic profile in patients with cardiovascular disease. The investigators hypothesize that a whole-food plant-based vegan diet will reduce markers of inflammation and improve glucometabolic profile compared with the American Heart Association (AHA)- recommended diet at 2 months follow-up in patients with coronary artery disease (CAD). The investigators are also evaluating endothelial function using the EndoPAT device and stool microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Subjects on stable medical therapy for at least 7-10 days post-coronary angiography and found to have CAD (defined as >50% lesion in an artery with >2mm caliber) .

Exclusion Criteria:

* Failure of the Treatment Self-Regulation Questionnaire
* Use of steroids or non-steroidal anti-inflammatory medications other than aspirin
* Use of probiotics or over the counter supplements other than standard vitamins
* Have a history of myocardial infarction or active infection within the preceding 3 months
* Have a history of an eating disorder or colon cleansing or are already on a whole-food plant-based vegan diet
* Have a planned PCI during the study period
* Are participating in a competing study
* Have any condition or situation that, in the investigator's opinion, may confound the study results, or may interfere significantly with the patient's ability to adhere with study procedures

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-03-11 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
change in hsCRP from baseline | At 8 weeks follow-up

SECONDARY OUTCOMES:
change in L-selectin from baseline | 4 week and 8 week follow-up
change in body mass index from baseline | 4 week and 8 week follow-up
change in Abdominal Circumference from baseline | 4 week and 8 week follow-up
change in Blood Pressure from baseline | 4 week and 8 week follow-up
change in CD11b from baseline | 4 week and 8 week follow-up
change in Stool microbiome from baseline | 4 and 8 week follow-up
change in EndPAT score from baseline | 4 and 8 week follow-up
change in Serum amyloid A from baseline | 4 week and 8 week follow-up
  soluble inflammatory marker
change in TNF-α from baseline | 4 week and 8 week follow-up
change in pentraxin-3 from baseline | 4 week and 8 week follow-up
change in MMP-9 from baseline | 4 week and 8 week follow-up
change in lipid panel from baseline | 4 week and 8 week follow-up
change in apolipoprotein B from baseline | 4 week and 8 week follow-up
change in fasting blood glucose from baseline | 4 week and 8 week follow-up
change in blood insulin from baseline | 4 week and 8 week follow-up
change in Hemoglobin a1c from baseline | 4 week and 8 week follow-up
change in cell adhesion molecule from baseline | 4 week and 8 week follow-up
change in monocyte subtype from baseline | 4 week and 8 week follow-up
change in interleukin from baseline | 4 week and 8 week follow-up
change in chemokine from baseline | 4 week and 8 week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Binita Shah, MD, MS, Principal Investigator — NYU SOM
Locations (1):
- NYUMC Tisch Hospital, HCC 14, New York, New York, United States